CLINICAL TRIAL: NCT05167942
Title: Exploration of the Deep Transcranial Magnetic Stimulation for Treatment Resistant Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20y11906300
Record Dates: First submitted 2021-12-10; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Treatment Resistant Schizophrenia Based on the DTMS
Keywords: Deep Transcranial Magnetic Stimulation; Treatment Resistant Schizophrenia; H1 coil
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham dTMS (Sham Comparator): 29 patients will be randomly allocated into this group,they will receive sham stimulation.
  Interventions: Device: deep transcranial magnetic stimulation with H1 coil
- dTMS 20Hz (Active Comparator): 29 patients will be randomly allocated into this group,they will receive real stimulation.
  Interventions: Device: High frequency deep transcranial magnetic stimulation with H1 coil
- dTMS iTBS (Active Comparator): 29 patients will be randomly allocated into this group,they will receive real stimulation.
  Interventions: Device: iTBS deep transcranial magnetic stimulation with H1 coil

INTERVENTIONS:
Device: deep transcranial magnetic stimulation with H1 coil — Sham deep transcranial magnetic stimulation on PFC .Duration:40 days.
  Arms: Sham dTMS
Device: High frequency deep transcranial magnetic stimulation with H1 coil — high frequency(20Hz) deep transcranial magnetic stimulation on PFC .Duration:40 days.
  Arms: dTMS 20Hz
Device: iTBS deep transcranial magnetic stimulation with H1 coil — iTBS deep transcranial magnetic stimulation on PFC .Duration:40 days.
  Arms: dTMS iTBS

SUMMARY:
Negative symptoms and cognitive dysfunction are of importance for the prognosis of the patients of schizophrenia. Based on the hypothesis that deep transcranial magnetic stimulation(dTMS) on prefrontal cortex #PFC# could down-regulate the glutamate level of PFC and regulate the functional network in patients with treatment resistance schizophrenia,this research plan to utilise multimodal functional magnetic imaging method(including structural MRI,resting-state functional magnetic resonance imaging and 1H-MRS) to investigate therapeutic efficacy of high-frequency deep transcranial magnetic stimulation on SZ patients symptoms,as well as to elucidate the correlation between treatment effects and glutamate level of PFC

DETAILED DESCRIPTION:
This study includes 87 treatment resistance schizophrenia patients. This study will investigate 1)abnormalities of the glutamate level of PFC in patients with schizophrenia compared to healthy controls by using 1H-MRS technique. 2)potential modulation effects of deep transcranial magnetic stimulation(dTMS) on prefrontal cortex function of patients with schizophrenia. 3)the therapeutic efficacy of dTMS on cognitive impairments and other psychotic symptoms of patients with schizophrenia by adopting cognitive function and psychotic symptoms evaluation,as well as to explore the optimal dTMS treatment pattern on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia who meet the dsm-5 diagnostic criteria
* Aged from 18 to 55
* Right-handedness, normal hearing, visual acuity or corrected visual acuity
* Written informed consent of the patient and his/her family
* All patients received MINI 7.0 structured interviews

Exclusion Criteria:

* Patients who are currently taking clozapine or who have failed to respond to a full course of treatment with clozapine
* Current or past neurological illness,severe physical illness,substance abuse or addiction,alcohol dependence,mental retardation,pregnancy or lactation,extreme agitation, stupor, negative suicide,or those who can not cooperate
* Medically unstable for at least 1 month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale(PANSS) | baseline,24 hours after the dTMS treatment,40 days
  Change from baseline in Positive and Negative Syndrome Scale(PANSS) after dtms treat 40 days
Change from baseline in MATRICS Consensus Cognitive Battery | baseline,24 hours after the rTMS treatment,40 days
  MATRICS Consensus Cognitive Battery

SECONDARY OUTCOMES:
Change of PFC neurogenesis | baseline,24 hours after the dTMS treatment,40days
  Quantify neural stem cells in hippocampal by using H1-MRS

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China